CLINICAL TRIAL: NCT04896424
Title: Does Vagal Response Indicate Cardiac Autonomic Modulation and Improve the Therapeutic Effect of Pulmonary Vein Isolation in Patients With Paroxysmal Atrial Fibrillation? Insides From Cryoballoon Ablation
Brief Title: Vagal Response and Cardiac Autonomic Modulation. Insides From Cryoballoon Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Radoslaw Kiedrowicz, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB-0012/91/10/15
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Vagal Nerve Stimulation; Autonomic Nervous System; Catheter Ablation
Keywords: atrial fibrillation; cardiac autonomic nervous system; cryoballoon ablation; ganglionated plexi; heart rate variability; vagal response
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryoballoon-based pulmonary veins isolation cohort (Other): Patients treated with a 28-mm second-generation cryoballoon (Arctic Front Advance, Medtronic) for paroxysmal atrial fibrillation and screened over a 2-year post-ablation period.
  Interventions: Procedure: cryoballoon-based pulmonary veins isolation

INTERVENTIONS:
Procedure: cryoballoon-based pulmonary veins isolation — A cryoballoon is introduced to the LA via a steerable sheath following a single transseptal puncture. The balloon is advanced toward the PV ostium and inflated. PV occlusion is documented by the injection of contrast. Optimal vessel occlusion is assumed when the PV showes complete contrast retention without any backflow to the atrium. The freezing time is chosen between 180 and 240s and left at the operator's discretion, along with a decision if to follow with a bonus-freeze cycle. The application is aborted and the cryoballoon is repositioned in the case of ineffective cooling or when the nadir temperature decreases < -60°C, to avoid excessive cooling. In cases where a real-time recording of PV potentials is available a short time-to-isolation<60s resultes in a single 180s freeze cycle. CBA always startes from the left upper PV (LUPV) followed by the left lower PV (LLPV).

SUMMARY:
The investigators sought to evaluate the incidence and influence of vagal response observed during cryoballoon-based pulmonary vein isolation on the cardiac autonomic nervous system (CANS) and ablation outcomes in paroxysmal atrial fibrillation cohort. 296 patients were treated with a 28-mm second-generation cryoballoon (Arctic Front Advance, Medtronic). Preprocedural pulmonary veins anatomy and their ostial dimensions were acquired with a computed tomography. 74 patients without structural heart disease and with no concomitant diseases were chosen for a detailed CANS assessment with heart rate variability analysis. All patients were screened over a 2-year post-ablation period.

DETAILED DESCRIPTION:
An interplay between left atrial (LA) ganglionated plexi (GP), a part of the intrinsic cardiac autonomic nervous system (CANS), and pulmonary veins (PVs) is considered to be an important mechanism related with the initiation and maintenance of atrial fibrillation (AF). Therefore additional GP ablation has been reported with better ablation outcomes when added to RF-based PV isolation (PVI). A cryoballoon ablation (CBA) is an anatomically based approach which allows PVI that is highly safe and efficacious. The extension of the scar created by the cryoballoon frequently extends beyond the PV orifice in the acute and chronic post-ablation phase creating a set of lesions that are near the LA-GP area and inadvertent damage. A marked vagal response (VR) observed during CBA is considered a marker for the CANS modification. However, changes in the autonomic tone were independently noted from the presence of VR in several studies. Moreover, it is not clear if these changes are transient or long-lasting, and it has been shown that the presence of VR increases ablation success although with conflicting results. In previous studies assessing the influence of CBA on the autonomic balance, CANS modulation was appraised with different surrogates, a small number of individuals were usually recruited and both paroxysmal and persistent AF populations were included. Therefore, the investigators sought to evaluate the incidence of VR observed during CBA-based PVI, its impact on CANS assessed with widely accepted heart rate variability (HRV) analysis, and in relation to ablation outcomes in a large paroxysmal AF (PAF) cohort.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of paroxysmal atrial fibrillation

Exclusion Criteria:

* Previous atrial fibrillation ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The number of patients free from atrial fibrillation following a cryoballoon-based pulmonary veins isolation beyond a 3-month blanking period. | 3 months
  Outpatient visit was scheduled at 3 months following ablation. A detailed medical history was taken with emphasis on registered atrial fibrillation episodes or atrial fibrillation suggestive symptoms. 24 hour Holter monitoring was performed in all patients.
The number of patients free from atrial fibrillation following a cryoballoon-based pulmonary veins isolation beyond a 3-month blanking period. | 6 months
  Outpatient visit was scheduled at 6 months following ablation. A detailed medical history was taken with emphasis on registered atrial fibrillation episodes or atrial fibrillation suggestive symptoms. 24 hour Holter monitoring was performed in all patients.
The number of patients free from atrial fibrillation following a cryoballoon-based pulmonary veins isolation beyond a 3-month blanking period. | 12 months
  Outpatient visit was scheduled at 12 months following ablation. A detailed medical history was taken with emphasis on registered atrial fibrillation episodes or atrial fibrillation suggestive symptoms. 24 hour Holter monitoring was performed in all patients.
The number of patients free from atrial fibrillation following a cryoballoon-based pulmonary veins isolation beyond a 3-month blanking period. | 18 months
  Outpatient visit was scheduled at 18 months following ablation. A detailed medical history was taken with emphasis on registered atrial fibrillation episodes or atrial fibrillation suggestive symptoms. 24 hour Holter monitoring was performed in all patients.
The number of patients free from atrial fibrillation following a cryoballoon-based pulmonary veins isolation beyond a 3-month blanking period. | 24 months
  Outpatient visit was scheduled at 24 months following ablation. A detailed medical history was taken with emphasis on registered atrial fibrillation episodes or atrial fibrillation suggestive symptoms. 24 hour Holter monitoring was performed in all patients.

OTHER OUTCOMES:
The incidence of vagal response observed during cryoballoon-based pulmonary veins isolation | At the time of procedure
  Vagal reaction was defined as sinus bradycardia <40 bpm, sinus arrest, atrioventricular block or hypotension registered anytime from the beginning of cryoapplication up to 1 minute following balloon deflation preceded by a thawing period.
The impact on of vagal response on intrinsic cardiac autonomic nervous system with widely accepted heart rate variability (HRV) analysis | 3 months
  A 24h holter ECG was acquired on the day before ablation and 3 months thereafter. Holter electrocardiograms were recorded by a DMS 300-3A (DM Software Inc., USA). A HRV was analysed by a Cardioscan II system (DM Software). Artifacts, premature complexes, and atrial runs were excluded from calculation. Records with abnormal beats, rhythms and noise that constituted >5% of all beats were repeated. HRV parameters included mean heart rate (mHR), five time-domain variables:(1) SDNN, (2) SDNN index, (3) SDANN, (4) rMSSD, (5) pNN50, and three frequency domain variables: (1) LF, (2) HF, and (3) LF/HF ratio
The impact on of vagal response on intrinsic cardiac autonomic nervous system with widely accepted heart rate variability (HRV) analysis | 6 months
  A 24h holter ECG was acquired on the day before ablation and 6 months thereafter. Holter electrocardiograms were recorded by a DMS 300-3A (DM Software Inc., USA). A HRV was analysed by a Cardioscan II system (DM Software). Artifacts, premature complexes, and atrial runs were excluded from calculation. Records with abnormal beats, rhythms and noise that constituted >5% of all beats were repeated. HRV parameters included mean heart rate (mHR), five time-domain variables:(1) SDNN, (2) SDNN index, (3) SDANN, (4) rMSSD, (5) pNN50, and three frequency domain variables: (1) LF, (2) HF, and (3) LF/HF ratio
The impact on of vagal response on intrinsic cardiac autonomic nervous system with widely accepted heart rate variability (HRV) analysis | 12 months
  A 24h holter ECG was acquired on the day before ablation and 12 months thereafter. Holter electrocardiograms were recorded by a DMS 300-3A (DM Software Inc., USA). A HRV was analysed by a Cardioscan II system (DM Software). Artifacts, premature complexes, and atrial runs were excluded from calculation. Records with abnormal beats, rhythms and noise that constituted >5% of all beats were repeated. HRV parameters included mean heart rate (mHR), five time-domain variables:(1) SDNN, (2) SDNN index, (3) SDANN, (4) rMSSD, (5) pNN50, and three frequency domain variables: (1) LF, (2) HF, and (3) LF/HF ratio

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw M Kiedrowicz, PhD, Principal Investigator — Pomeranian Medical University

IPD SHARING:
Plan to Share IPD: No